CLINICAL TRIAL: NCT04016974
Title: A Multiple-dose, Single-centre, Randomised, Double-blind, Placebo-controlled Trial to Investigate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Oral Semaglutide in Healthy Chinese Subjects
Brief Title: A Research Study of How Oral Semaglutide Tablets Work in Healthy People Who Are Chinese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9924-4303; U1111-1186-6753 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteers; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral semaglutide (Experimental)
  Interventions: Drug: Oral semaglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral semaglutide — Semaglutide tablets once daily as follows: 3 mg for the first treatment period (day 1-28), followed by 7 mg in the second treatment period (day 29-56), followed by 14 mg in the third treatment period (day 57-84)
  Arms: Oral semaglutide
Drug: Placebo — Placebo tablets once daily throughout the treatment period (day 1 to 84)
  Arms: Placebo

SUMMARY:
This study looks at the way a new medicine tablet called semaglutide moves in and throughout the body over time. It will also look at if the medicine is safe and the body can accept it. The new medicine is planned to treat diabetes. The aim of the study is to see how semaglutide tablets work in healthy people who are Chinese. Participants will either get oral semaglutide tablets or placebo (dummy) tablets - which treatment is decided by chance. The tablet form of semaglutide is a new medicine that cannot be prescribed. Doctors can prescribe semaglutide as an injection only. It is for the treatment of diabetes in some countries. Participants will get 1 tablet per day for 12 weeks (84 days). Participants will get 1 tablet a day to take with up to half a glass of water (maximum 120 mL). Participants must take the tablet first thing in the morning on an empty stomach (water is allowed until 2 hours before taking the tablet). After taking the tablet, participants must not eat or drink anything for at least 30 minutes. After 30 minutes, they can have their first meal of the day and take any other medicines they may need, such as birth control tablets, routine vitamins and use of paracetamol at times.

ELIGIBILITY:
Inclusion Criteria:

* Chinese male or female, aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body weight equal to or above 54.0 kg
* Body mass index (BMI) between 20.0 and 24.9 kg/m^2 (both inclusive)
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, ECG and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using highly effective contraceptive methods
* History of pancreatitis (acute or chronic) as declared by the subject.
* Family or personal history of multiple endocrine neoplasia type 2 (MEN2) or medullary thyroid carcinoma (MTC) as declared by the subject.
* History or presence of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer and in-situ carcinomas) as declared by the subject.
* History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g., subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery) as declared by the subject.
* Smoker (defined as a subject who is smoking equal to or more than 1 cigarette or the equivalent per day).
* Unable or unwilling to refrain from smoking and use of nicotine substitute products during the inpatient periods, as judged by the investigator.
* Any blood draw in excess of 25 mL in the past month, or donation of blood or plasma in excess of 400 mL within the 3 months preceding screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-01-23 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
AUC0-24h,sema,SS, area under the semaglutide concentration-time curve during a dosing interval (0-24 hours) at steady state | After the last dose of oral semaglutide at dose levels of 3 mg on day 28 and 7 mg on day 56, and after the last 3 daily doses of oral semaglutide at dose level 14 mg on day 82, 83 and 84
  h*nmol/L

SECONDARY OUTCOMES:
Cmax,sema,SS, maximum observed semaglutide plasma concentration during a dosing interval (0-24 hours) at steady state | After the last dose of oral semaglutide at dose levels of 3 mg on day 28 and 7 mg on day 56, and after the last 3 daily doses of oral semaglutide at dose level 14 mg on day 82, 83 and 84
  nmol/L
tmax,sema,SS, time to maximum observed semaglutide plasma concentration during a dosing interval (0-24 hours) at steady state | After the last dose of oral semaglutide at dose levels of 3 mg on day 28 and 7 mg on day 56, and after the last 3 daily doses of oral semaglutide at dose level 14 mg on day 82, 83 and 84
  h
CL/Fsema,SS, total apparent clearance of semaglutide at steady state | After the last dose of oral semaglutide at dose levels of 3 mg on day 28 and 7 mg on day 56, and after the last 3 daily doses of oral semaglutide at dose level 14 mg on day 82, 83 and 84
  L/h
Ctrough,sema,SS, trough semaglutide plasma concentration at steady state | After the last 3 daily doses of oral semaglutide administration at 3, 7 and 14 mg dose levels on day 27-29, 55-57 and 83-85
  nmol/L
t½,sema,SS, terminal half-life of semaglutide at steady state | After the last dose of oral semaglutide 14 mg on day 84
  h
Vss/Fsema, apparent volume of distribution of semaglutide at steady state | After the last dose of oral semaglutide 14 mg on day 84
  L
MRTsema,SS, mean residence time of semaglutide at steady state | After the last dose of oral semaglutide 14 mg on day 84
  h
Rtheor,sema,SS, theoretical accumulation index, which is defined as [1/(1-Exp (-λZ,sema,SS*24h))], where λZ,sema,SS=log(2)/t½,sema,SS | After the last dose of oral semaglutide 14 mg on day 84
  Index value
Change in body weight from baseline | Day 1, day 85
  kg
Change in fasting plasma glucose from baseline | Day 1, day 85
  mmol/l
Number of treatment-emergent adverse events | From the time of first dosing (day 1) until completion of the follow-up visit (day 119-121)
  Count
Number of treatment-emergent hypoglycaemic episodes | From the time of first dosing (day 1) until completion of the follow-up visit (day 119-121)
  Count

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Beijing Hospital-phase I, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Xie P, Abildlund MT, Baekdal TA, He X, Lyauk YK, Patted URH, Ning Z, Shi A. A phase 1, randomized, double-blind, placebo-controlled trial investigating the pharmacokinetics, pharmacodynamics, safety and tolerability of oral semaglutide in healthy Chinese subjects. Diabetes Obes Metab. 2024 Aug;26(8):3068-3077. doi: 10.1111/dom.15624. Epub 2024 May 29. PMID 38808476